CLINICAL TRIAL: NCT04956653
Title: An Analysis of Social Characteristics of Hospitalized Patients With Spinal Degenerative Diseases in the Orthopedic Department of Peking University Third Hospital During 2003-2016
Brief Title: Social Characteristics of Hospitalized Patients With Spinal Degenerative Diseases
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018082
Record Dates: First submitted 2021-07-02; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Spinal Degenerative Diseases
Keywords: Spinal Degenerative Diseases; social characteristics; hospitalized patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients diagnosed with Cervical Degenerative Disease: Patients who suffered from Cervical Degenerative Disease, treated by operation for the first time and aged 18 years old or over were assigned to CDD group.
  Interventions: Other: Without additional intervention
- Patients diagnosed with Thoracic Degenerative Disease: Patients who suffered from Thoracic Degenerative Disease, treated by operation for the first time and aged 18 years old or over were assigned to TDD group.
  Interventions: Other: Without additional intervention
- Patients diagnosed with Lumbar Degenerative Disease: Patients who suffered from Lumbar Degenerative Disease, treated by operation for the first time and aged 18 years old or over were assigned to LDD group.
  Interventions: Other: Without additional intervention

INTERVENTIONS:
Other: Without additional intervention — Only patients' information was collected

SUMMARY:
To explore the correlation of the incidence and social characteristics in patients with spinal degenerative diseases (SDD), and to provide certain evidence for prevention, treatment and incidence control of the disease.

DETAILED DESCRIPTION:
Objectives: To explore the correlation of the incidence and social characteristics in patients withspinal degenerative diseases (SDD), and to provide certain evidence for prevention, treatment and incidencecontrol of the disease. Methods: Data between January 1, 2003 to December 31, 2016 were collected from electronic medical documents of the orthopedic department, including patients who suffered from SDD, treated by operation for the first time and aged 18 years old or over. Descriptive statistics and Chi-square test were used to analyze the correlation of social characteristics of patients（eg. age, gender, career, place of birth, nationality and comorbidities）and the degenerative spinal diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as spinal disc herniation (prolapse), spinal stenosis, Non-traumatic spinal instability, spondylolisthesis, degenerative scoliosis not caused by congenital spinal deformity. 2. Hospitalized patients under operation. 3. Over 18 yrs. 4. Patients in North China.

Exclusion Criteria:

- Patients diagnosed as Hypertrophy of Posterior Longitudinal Ligament or Hypertrophy of Ligamentum Flavum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 32522 surgical inpatients were selected from Peking University Third Hospital during 2003-2016.
Sampling Method: Non-Probability Sample
Enrollment: 32502 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Population characteristics of hospitalized patients | 2003-2016
  Correlation analysis of population characteristics and spinal degenerative diseases (SDD)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No